CLINICAL TRIAL: NCT00614770
Title: A Multicenter, Prospective, Randomized Controlled Trial for the Detection of Colon Polyps and Predicting Histology
Brief Title: Narrow Band Imaging Colon Polyp Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); Midwest Biomedical Research Foundation (Other)
Responsible Party: Amit Rastogi, MD, Kansas City VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AR0003; AR0003
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Adenomatous Polyp; New Imaging Techniques in Colonoscopy
Keywords: colonoscopy
MeSH Terms: conditions — Adenomatous Polyps | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Standard White Light Colonoscopy
  Interventions: Procedure: standard of care colonoscopy
- 2 (Experimental): High Definition White Light Colonoscopy
  Interventions: Procedure: standard of care colonoscopy
- 3 (Experimental): Narrow Band Imaging Colonoscopy
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: standard of care colonoscopy — Standard White Light Colonoscopy
  one exam per patient
  Arms: 1
Procedure: colonoscopy — Narrow Band Imaging Colonoscopy
  one exam per patient
  Arms: 3
Procedure: standard of care colonoscopy — High Definition White Light Colonoscopy
  one exam per patient
  Arms: 2

SUMMARY:
In this study the investigators hypothesize that High Definition White Light colonoscopy and narrow band imaging (NBI) will detect a higher number of adenomas compared to standard definition white light colonoscopy. NBI will have a higher accuracy in predicting polyp histology compared to high definition colonoscopy and standard colonoscopy.

Specific Aim 1 - To compare the prevalence of adenomas detected by standard colonoscopy, high-definition white light colonoscopy and NBI.

Specific Aim 2 - To compare the number of adenoma detected per subject by standard colonoscopy, high-definition white light colonoscopy and NBI.

Specific Aim 3 - To compare the accuracy of predicting polyp histology between standard colonoscopy, high-definition white light colonoscopy and NBI by evaluating the surface mucosal and vascular patterns during the procedure.

Specific Aim 4 - To determine the inter-observer agreement between investigators for the recognition of various polyp patterns

DETAILED DESCRIPTION:
This study is a multi-center randomized controlled trial that will be conducted at the Kansas City VA Medical Center, Kansas City, MO and The Barnes Jewish Hospital, St Louis, MO. Patients referred for screening and surveillance colonoscopy will be enrolled. They will be randomized to one of the following three groups: standard white light colonoscopy, high-definition white light colonoscopy or NBI.

All colonoscopies will be performed at the Kansas City VA Medical Center and The Barnes Jewish Hospital, St Louis, MO. Moderate sedation will be administered for the procedure with intravenous midazolam, demerol or fentanyl and Propofol. In patients randomized to the NBI arm, the colonoscope will be inserted to the cecum under white light and will switch to NBI mode at the time of withdrawal. After cecal intubation, the colonic mucosa will be carefully visualized during withdrawal of the scope with one of the three imaging modalities to which the patient has been randomized. No effort will be made to look for polyps during the insertion of the colonoscope. All polyps detected will be documented for their size, morphology (Polypoid: sessile, pedunculated or Non polypoid: superficially elevated, completely flat, depressed), and location. The surface of the polyp will be assessed during the procedure and the histology will be predicted real time by evaluating the surface mucosal and vascular patterns. The patterns would be classified into one of the four patterns described in our pilot study (tubular and gyrus patterns will be combined to tubulogyrus pattern). Any other patterns detected would be described and kept in the miscellaneous category. If a pattern is not identified on a polyp with either white light or NBI, it will be recorded as such and no attempts will be made to predict histology. Photo documentation of the surface patterns of the polyps will be performed. Polyps will then be removed either with a biopsy forcep or snare and sent for histopathological evaluation. Each polyp removed will have one or more corresponding picture of its surface patterns and these will be labeled accordingly. The total time spent in inspecting the colonic mucosa (excluding the time spent in removal of polyps or clearing the colon of liquid and solid debris) will be measured with a stop watch. Representative images of the various polyp patterns will be reviewed, discussed and standardized amongst all the investigators at both sites. In addition, images of all the polyp patterns will be printed and posted in the endoscopy suites at both hospitals.

The bowel preparation will be evaluated and graded as follow:

Excellent (score=1) - >90% mucosa seen, mostly liquid colonic contents, minimal suctioning needed for adequate visualization.

Good (score=2) - >90% of mucosa seen, mostly liquid colonic contents, significant suctioning needed for adequate visualization Fair (score=3) - > 90% mucosa seen, mixture of liquid and semisolid colonic contents, could be suctioned and/or washed Inadequate (score=4) - <90% mucosa seen, mixture of semisolid ands solid colonic contents, which could not be suctioned or washed

Patients with "Inadequate" (score = 4) bowel prep will be excluded.

ELIGIBILITY:
Inclusion criteria:

* referral for screening or surveillance colonoscopy
* the ability to provide informed consent

Exclusion criteria:

* prior surgical resection of any portion of colon
* prior history of colon cancer
* history of inflammatory bowel disease
* use of anti-platelet agents or anticoagulants that precludes removal of polyps during the procedure
* poor general condition or any other reason to avoid prolonged procedure time
* history of polyposis syndrome or HNPCC
* inability to give informed consent.
* Inadequate bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2008-02; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The prevalence of adenomas in the three arms of the study. | 2 years
  Number of subjects with adenomas in the three arms of the study

SECONDARY OUTCOMES:
Secondary outcome will be number of adenomas detected per subject in the three arms, the sensitivity, specificity, and accuracy of predicting polyp histology real time by the three imaging modalities. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Rastogi, MD, Principal Investigator — Kansas City VA Medical Center
Locations (2):
- United States (2):
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri

REFERENCES:
- [Derived] Rastogi A, Early DS, Gupta N, Bansal A, Singh V, Ansstas M, Jonnalagadda SS, Hovis CE, Gaddam S, Wani SB, Edmundowicz SA, Sharma P. Randomized, controlled trial of standard-definition white-light, high-definition white-light, and narrow-band imaging colonoscopy for the detection of colon polyps and prediction of polyp histology. Gastrointest Endosc. 2011 Sep;74(3):593-602. doi: 10.1016/j.gie.2011.04.050. Epub 2011 Jul 29. PMID 21802078